CLINICAL TRIAL: NCT01811615
Title: A Clinical Study to Investigate the Efficacy of New Alcohol Free Mouthrinses
Brief Title: Efficacy of New Alcohol Free Mouthrinses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, PD Dr. A. Rainer Jordan, Head of Section Preclinical Dentistry, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OHCMA-CHM-BUH-RHS-00633
Record Dates: First submitted 2013-01-18; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Gum Disease
MeSH Terms: conditions — Gingival Diseases | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- toothbrushing plus rinsing (Active Comparator): 0.06% CHX + 0.025% NaF plus toothbrushing and alcohol-containing mouth rinsing
  Interventions: Other: alcohol-containing mouth rinsing
- alcohol-free experimental mouth rinse (Experimental): 0.06% CHX + 0.025% NaF plus toothbrushing
  Interventions: Other: alcohol-free experimental mouth rinse
- toothbrushing and rinsing (Experimental): 0.06% CHX + 0.03% CPC + 0.025% NaF, alcohol-free, mouth rinsing
  Interventions: Other: alcohol-free experimental mouth rinse
- toothbrushing alone (No Intervention): negative control

INTERVENTIONS:
Other: alcohol-free experimental mouth rinse
  Arms: alcohol-free experimental mouth rinse; toothbrushing and rinsing
Other: alcohol-containing mouth rinsing
  Arms: toothbrushing plus rinsing

SUMMARY:
Background To evaluate the efficacy of two alcohol-free antimicrobial mouthrinses in reducing plaque and gingivitis compared to an alcohol-containing rinse and toothbrushing alone.

Methods 160 healthy volunteers were enrolled in the parallel-design examiner-blind study. After screening and stratification by sex and papillary bleeding index (PBI), participants were randomly and equally assigned to four groups: (1) toothbrushing + rinsing (0.06% CHX + 0.025% NaF, alcohol-containing rinse, Corsodyl® Daily Defence Mouthwash; positive control); (2) toothbrushing + rinsing (0.06% CHX + 0.025% NaF, alcohol-free experimental rinse); (3) toothbrushing + rinsing (0.06% CHX + 0.03% CPC + 0.025% NaF, alcohol-free experimental rinse); (4) toothbrushing alone (negative control). At baseline, Quigley-Hein plaque index (QHI), the modified proximal plaque index (MPPI), and PBI were recorded. All subjects were advised to brush their teeth as usual during the eight weeks study period. Additionally, groups 1-3 were instructed to rinse twice daily (30 sec. each). All participants used Dr. Best multi aktiv toothpaste and Dr. Best plus toothbrush (medium stiffness). Eight weeks after baseline, indices were recorded again. Anova with Bonferroni adjustment was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* participants between 18 and 65 years
* no severe periodontitis
* informed consent

Exclusion Criteria:

* handicapped participants
* allergies against mouth rinses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Modified Proximal Plaque Index (MPPI) | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zimmer, Professor, Study Director — Witten/Herdecke University
Locations (1):
- Witten/Herdecke University School of Dental Medicine, Witten, North Rhine-Westphalia, Germany